CLINICAL TRIAL: NCT02582840
Title: A Clinical Pharmacology and Long Term Study to Evaluate the Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of Dapagliflozin Therapy in Combination With Insulin in Japanese Subjects With Type 1 Diabetes Who Have Inadequate Glycemic Control
Brief Title: The PK and PD of Dapagliflozin Therapy in Combination With Insulin in Japanese Subjects With T1DM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D1695C00001sub
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Results first posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2018-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Japanese patients with type 1 diabetes with inadequate glycemic control on insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- dapagliflozin 5mg (Experimental): dapagliflozin tablet 5mg
  Interventions: Drug: Dapagliflozin 5mg
- dapagliflozin 10mg (Experimental): dapagliflozin tablet 10mg
  Interventions: Drug: Dapagliflozin 10mg
- Placebo (Placebo Comparator): dapagliflozin tablet 5mg placebo or 10 mg placebo
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: Dapagliflozin 5mg — Dapagliflozin, a blood glucose lowering drug. Oral dose
  Arms: dapagliflozin 5mg
Drug: Dapagliflozin 10mg — Dapagliflozin, a blood glucose lowering drug. Oral dose
  Arms: dapagliflozin 10mg
Drug: Placebo tablet — Placebo tablet. Oral dose
  Arms: Placebo

SUMMARY:
This randomized, single-blind, 3 arm, parallel group, placebo controlled PK/PD study will enrol 30 Japanese male and female patients with T1DM and age 18 to 65 years, with inadequate glycemic control on insulin defined as HbA1c ≥ 7.0% and ≤ 10.0% at screening visit. lacebo-controlled design. Patients will be randomized in a 1:1:1 ratio into one of the 3 single-blinded treatment arms; dapagliflozin 5 mg, dapagliflozin 10 mg or placebo. CSII user are excluded.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent Subjects or their legally responsible representatives must be willing and able to give signed and dated written informed consent.
* Target Population Diagnosis of T1DM. In addition, the following criteria also needs to be met; Central laboratory test of C-peptide < 0.7 ng/mL Subject re-enrolment: This study does not permit the re-enrolment of a subject who has discontinued the study as a screen failure
* Insulin use for at least 12 months prior to the enrolment per subject report or medical records and Method of insulin administration (MDI) must have been unchanged for at least 3 months prior to the enrolment per subject report or medical records. Subjects must be taking a total daily insulin dose of ≥ 0.3 U/kg/day for at least 3 months prior to the enrolment. CSII users are excluded. MDI insulin administration subject must be on ≥ 3x injections per day.
* Gender and reproductive Status Japanese men and women.
* HbA1c eligibility criteria include: Screening Visit: Central laboratory HbA1c ≥ 7.0 % and ≤ 10.0 % (One repeat HbA1c test for subjects in screening if their initial test result was an HbA1c ± 0.2% of the cut off values)
* BMI ≥ 20.0 kg/m², ≤ 35.0 kg/m² at visit 1
* Ages 18 to 65 years, inclusive - ≥ 18 years old and < 20 years old must have assent forms signed and dated by their parents or guardians

Exclusion Criteria:

* Target Disease Exceptions History of T2DM In cases where the subject has a history of T2DM and has a documented history of being auto-antibody positive for GAD65, tyrosine phosphatase IA-2/IA-2β, or Zinc Transporter 8 (ZnT8), or fasting c-peptide value below the lower limit of detection performed by local or central laborator, the subject will be eligible for screening
* Maturity onset diabetes of young (MODY), Pancreatic surgery, chronic pancreatitis, or other pancreatic disorders that could result in decreased β-cell capacity (eg, pancreatogenous diabetes)
* Any antihyperglycemic agent use, other than thiazolidinediones, or insulin, within 1 month prior to the screening visit. Use of thiazolidinediones within 6 months prior to the screening visit.
* History of DKA requiring medical intervention (eg, emergency room visit and/or hospitalization) within 1 month prior to the enrolment
* History of hospital admission for glycemic control (either hyperglycemia or hypoglycemia) within 1 month prior to the enrolment
* Malignancy within 5 years of the enrolment (with the exception of treated basal cell or treated squamous cell carcinoma)
* History of bladder cancer
* History of radiation therapy to the lower abdomen or pelvis at any time Unstable pre-proliferative and proliferative retinopathy (untreated or under treatment).
* Physical and Laboratory Test Findings Aspartate aminotransferase (AST) > 3x upper limit of normal (ULN) Alanine aminotransferase (ALT) > 3x ULN Serum total bilirubin (TB) > 2.0 mg/dL (34.2 μmol/L).
* Estimated GFR (eGFR) by the Japanese Society of Nephrology formula ≤ 60 mL/min/1.73m2. Hemoglobin ≤ 11.0 g/dL (110 g/L) for men; hemoglobin ≤ 10.0 g/dL (100 g/L) for women.
* Positive for hepatitis B surface antigen or anti-hepatitis C virus antibody
* Abnormal Free T4

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fukuoka, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 26 October 2015 to 04 June 2016, Japan, patients with type 1 diabetes mellitus.
Pre-assignment Details: Of 62 patients who signed informed consent, 42 eligible patients randomized and completed the 7-day treatment period (Part A) of the study.
Groups:
- Placebo + Insulin: Placebo administered orally once daily in the morning.
- Dapagliflozin 5mg + Insulin: Dapagliflozin 5 mg administered orally once daily in the morning.
- Dapagliflozin 10 mg + Insulin: Dapagliflozin 10 mg administered orally once daily in the morning.
Period: Overall Study
Arm/Group | Placebo + Insulin | Dapagliflozin 5mg + Insulin | Dapagliflozin 10 mg + Insulin
Started | 14 | 14 | 14
Completed | 14 | 14 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Insulin | Dapagliflozin 5mg + Insulin | Dapagliflozin 10 mg + Insulin | Total
Number analyzed (Participants) | 14 | 14 | 14 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (10.62) | 37.0 (10.05) | 37.1 (10.21) | 38.9 (10.38)
Age, Customized [Number; unit: Participants]
  <45 Years | 10 | 10 | 10 | 30
  >=45 Years | 4 | 4 | 4 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 7 | 24
  Male | 3 | 8 | 7 | 18
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 14 | 14 | 14 | 42
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 14 | 14 | 14 | 42
Duration of Type 1 Diabetes [Mean (Standard Deviation); unit: years] | 16.89 (10.530) | 15.94 (9.235) | 14.69 (12.368) | 15.84 (10.561)
Hemoglobin A1c (HbA1c)% [Mean (Standard Deviation); unit: percent of hemoglobin] | 8.13 (0.835) | 7.91 (0.610) | 7.89 (0.553) | 7.98 (0.669)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 134.00 (63.898) | 142.93 (49.930) | 133.36 (42.239) | 136.76 (51.675)
C-Peptide [Number; unit: Participants]
  < 0.1 ng/mL | 12 (0.083) | 13 (0.107) | 11 (0.036) | 0.12 (0.079)
  >= 0.1 ng/mL | 2 | 1 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Dapagliflozin Maximum Observed Plasma Concentration (Cmax) of 7 Days Repeated Doses of Dapagliflozin - Pharmacokinetic (PK) Set
Description: Serial blood samples for determination of study drug were collected predose Day 1, Day 7 (60 minutes prior to dose), Day 7 (0, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dose).
Time Frame: Day 1-7
Population: Pharmacokinetic set - Part A (PK-A): The PK set consisted of all randomized subjects who had at least one dose of randomized study medication for Part A and had an evaluable plasma concentration data of dapagliflozin and/or its major metabolite dapagliflozin 3-O-glucuronide.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Dapagliflozin 10mg + Insulin: Dapagliflozin 10 mg administered orally once daily in the morning.
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 10 | 10
ng/mL | 69.31 (26.42) | 162.09 (26.03)

2. Primary Outcome: Dapagliflozin Minimum Observed Plasma Concentration (Cmin) of 7 Days Repeated Doses of Dapagliflozin - Pharmacokinetic (PK) Set
Description: as for outcome 1
Time Frame: Day 1-7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 10 | 10
ng/mL | 3.40 (80.14) | 5.71 (52.36)

3. Primary Outcome: Dapagliflozin Time of Maximum Observed Plasma Concentration (Tmax) of 7 Days Repeated Doses of Dapagliflozin - Pharmacokinetic (PK) Set
Description: as for outcome 1
Time Frame: Day 1-7
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 10 | 10
hours | 2.00 (52.36) [1.00 to 3.00] | 2.00 [1.00 to 3.00]

4. Primary Outcome: Dapagliflozin Area Under the Concentration-time Curve From Time Zero to Time of the Last Quantifiable Concentration AUC(0-T) of 7 Days Repeated Doses of Dapagliflozin - Pharmacokinetic (PK) Set
Description: as for outcome 1
Time Frame: Day 1-7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 10 | 10
ng*h/mL | 322.72 (44.69) [1.00 to 3.00] | 670.01 (36.92)

5. Primary Outcome: Dapagliflozin 3-O-Glucuronide Maximum Observed Plasma Concentration (Cmax) of 7 Days Repeated Doses of Dapagliflozin - Pharmacokinetic (PK) Set
Description: as for outcome 1
Time Frame: Day 1-7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 10 | 10
ng/mL | 61.88 (31.95) | 136.62 (31.96)

6. Primary Outcome: Dapagliflozin 3-O-Glucuronide Minimum Observed Plasma Concentration (Cmin) of 7 Days Repeated Doses of Dapagliflozin - Pharmacokinetic (PK) Set
Description: as for outcome 1
Time Frame: Day 1-7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 10 | 10
ng/mL | 3.89 (56.43) | 6.25 (35.45)

7. Primary Outcome: Dapagliflozin 3-O-Glucuronide Time of Maximum Observed Plasma Concentration (Tmax) of 7 Days Repeated Doses of Dapagliflozin - Pharmacokinetic (PK) Set
Description: as for outcome 1
Time Frame: Day 1-7
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 10 | 10
hours | 2.00 (52.36) [1.00 to 4.00] | 2.00 [1.00 to 3.00]

8. Primary Outcome: Dapagliflozin 3-O-Glucuronide Area Under the Concentration-time Curve From Time Zero to Time of the Last Quantifiable Concentration AUC(0-T) of 7 Days Repeated Doses of Dapagliflozin - Pharmacokinetic (PK) Set
Description: as for outcome 1
Time Frame: Day 1-7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 10 | 10
ng*h/mL | 345.87 (29.32) [1.00 to 3.00] | 675.50 (23.66)

9. Primary Outcome: Dapagliflozin Ratio of Metabolite to Parent AUC of 7 Days Repeated Doses of Dapagliflozin - Pharmacokinetic (PK) Set
Description: as for outcome 1
Time Frame: Day 1-7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Dapagliflozin 5mg + Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 10 | 10
ratio | 0.75 (44.26) [1.00 to 3.00] | 0.70 (30.40)

10. Primary Outcome: 24-hour Urinary Glucose (g/24h) Mean Change From Baseline on Day 7 - Pharmacodynamic (PD) Set
Description: The 24-hour period is defined based on the morning void, from the first morning void to the one of the next day.
Time Frame: Baseline (the last available assessment prior to the first dose of study medication), Day 7
Population: Pharmacodynamic set Part A (PD-A): The PD set consisted of all randomized subjects who received at least one dose of randomized study medication for Part A, and who had a non missing baseline value and at least one post-baseline value for at least one pharmacodynamic variable.
Measure: Mean (Standard Deviation); unit: g/24-hour
Groups:
- Dapagliflozin 5mg+ Insulin: Dapagliflozin 5 mg administered orally once daily in the morning.
Arm/Group | Placebo + Insulin | Dapagliflozin 5mg+ Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 14 | 14 | 14
g/24-hour | -6.16 (30.337) [1.00 to 3.00] | 96.55 (30.083) | 101.28 (20.129)

11. Secondary Outcome: Total Daily Insulin (IU) Percent Change From Baseline to Day 7 - Pharmacodynamic (PD) Set
Description: Total daily insulin dose is defined as the sum of all insulin doses (basal+bolus+premixed) for each day. Mean percent change from baseline was calculated using the geometric mean back-transformed from the results calculated under the logarithm transformation.
Time Frame: Baseline (the last available assessment on or prior to the first dose of study medication), Day 7
Population: as for outcome 10
Measure: Mean (Standard Error); unit: percent chagne
Arm/Group | Placebo + Insulin | Dapagliflozin 5mg+ Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 14 | 14 | 14
percent chagne | -4.97 (5.280) [1.00 to 3.00] | -36.86 (3.324) | -39.13 (2.675)

12. Secondary Outcome: Daily Basal Insulin (IU) Percent Change From Baseline to Day 7 - Pharmacodynamic (PD) Set
Description: Mean percent change from baseline was calculated using the geometric mean back-transformed from the results calculated under the logarithm transformation.
Time Frame: Baseline (the last available assessment on or prior to the first dose of study medication), Day 7
Population: as for outcome 10
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo + Insulin | Dapagliflozin 5mg+ Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 14 | 14 | 14
percent change | -16.75 (7.215) [1.00 to 3.00] | -36.74 (5.671) | -39.63 (3.466)

13. Secondary Outcome: Daily Bolus Insulin (IU) Percent Change From Baseline to Day 7 - Pharmacodynamic (PD) Set
Description: as for outcome 12
Time Frame: Baseline (the last available assessment on or prior to the first dose of study medication), Day 7
Population: as for outcome 10
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo + Insulin | Dapagliflozin 5mg+ Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 14 | 14 | 14
percent change | 4.56 (5.905) [1.00 to 3.00] | -36.06 (4.238) | -39.89 (3.367)

14. Secondary Outcome: Fasting Plasma Glucose (FPG) (mg/dL) Change From Baseline to Day 7 - Pharmacodynamic (PD) Set
Time Frame: Baseline (the last available assessment on or prior to the first dose of study medication), Day 7
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo + Insulin | Dapagliflozin 5mg+ Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 14 | 14 | 14
mg/dL | 11.0 (41.31) [1.00 to 3.00] | -10.4 (62.10) | -13.1 (44.69)

15. Secondary Outcome: Seated Systolic Blood Pressure (mmHG) Change From Baseline to Day 7 - Pharmacodynamic (PD) Set
Time Frame: Baseline (the last available assessment on or prior to the first dose of study medication), Day 7
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Placebo + Insulin | Dapagliflozin 5mg+ Insulin | Dapagliflozin 10mg + Insulin
Number analyzed (Participants) | 14 | 14 | 14
mmHG | -3.1 (7.81) [1.00 to 3.00] | -2.1 (7.71) | 1.5 (10.66)

ADVERSE EVENTS:
Time Frame: Non-serious adverse event (AE): onset on or after the 1st day of dose up to on or prior to the last day of dose plus 4 days. Serious AE: onset on or after the 1st day of dose up to on or prior to the last day of dose plus 30 days.
Arm/Group | Placebo + Insulin | Dapagliflozin 5mg + Insulin | Dapagliflozin 10 mg + Insulin
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 2/14 | 5/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Insulin (N=14) | Dapagliflozin 5mg + Insulin (N=14) | Dapagliflozin 10 mg + Insulin (N=14)
THIRST (General disorders) | 0 (0) | 1 (1) | 4 (4)
MALAISE (General disorders) | 0 (0) | 0 (0) | 1 (1)
MUMPS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
URINE OUTPUT INCREASED (Investigations) | 0 (0) | 0 (0) | 2 (2)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other